CLINICAL TRIAL: NCT05667090
Title: Effects of Multiple Mega-dose of Vitamin D3 Supplementation on Ameliorating Moderate to Severe Chronic Pain in Hemodialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N202209072
Record Dates: First submitted 2022-12-18; First posted 2022-12-28 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-12

CONDITIONS: Hemodialysis; Chronic Pain; Hyperparathyroidism
Keywords: Vitamin D supplementation; Mega-dose vitamin D; Cholecalciferol; Chronic pain
MeSH Terms: conditions — Chronic Pain; Hyperparathyroidism | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental): Oral supplementaiton of 2,304,000 IU vitamin D3 in 4 weeks
  Interventions: Other: Vitamin D
- Placebo Group (Placebo Comparator): Oral supplementaiton of placebo in 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vitamin D — Oral supplementaiton of 576,000 IU once a week of vitamin D3 for 4 weeks
  Arms: Vitamin D group
Other: Placebo — Oral supplementaiton of placebo once a week for 4 weeks
  Arms: Placebo Group

SUMMARY:
Pain is a major complaint in hemodialysis (HD) patients. Concentrations of parathyroid hormone (PTH) >250 pg/ml are associated with chronic pain. Visual Analogue Scale (VAS) score which is used to assess the pain severity is positively related to PTH levels. This study is aimed to assess the effects of multiple mega dosages vitamin D supplementations in HD patients with chronic pain. It's a single-center, parallel, double-blind randomized control trial that administrations of 576,000 IU once a week of vitamin D3 for 4 weeks or placebo are for 120 eligible subjects. VAS and laboratory tests including serum concentrations of 25(OH)D, calcium, phosphorus, PTH and C-reactive protein will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Haemodialysis subject ≥ 20 years old
2. iPTH > 250 pg/mL
3. Chronic pain with visual analogue scale (VAS) score ≥ 4
4. Voluntary to check serum 25(OH)D levels two times by his/her own payment during the study
5. Sign the informed consent

Exclusion Criteria:

1. Used to participate in other clinical trials
2. Chronic liver disease
3. Sarcoidosis or multiple myeloma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale of Pain | Baseline (day 1)
Visual Analogue Scale of Pain | week 2 (day 8)
Visual Analogue Scale of Pain | week 3 (day 15)
Visual Analogue Scale of Pain | week 4 (day 22)
Visual Analogue Scale of Pain | week 5 (day 29)

SECONDARY OUTCOMES:
25(OH)D level | Baseline (day 1) and week 5 (day 29) post-supplementation
Serum calcium | Baseline (day 1) and week 5 (day 29) post-supplementation
Serum phosphorus | Baseline (day 1) and week 5 (day 29) post-supplementation
C-reactive protein (CRP) test | Baseline (day 1) and week 5 (day 29) post-supplementation
Concentrations of parathyroid hormone (PTH) | Baseline (day 1) and week 5 (day 29) post-supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No